CLINICAL TRIAL: NCT02454439
Title: Assessment of Cardiac Resynchronization Therapy in Patients With Wide QRS and Non-specific Intraventricular Conduction Delay: a Randomized Trial
Acronym: NICD-CRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHU-0233; 2014-A01848-39 (Registry Identifier: 2014-A01848-39)
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2015-09

CONDITIONS: Heart Failure
Keywords: Heart Failure with reduced ejection fraction (<35%); Cardiac Resynchronisation Therapy; Non specific intraventricular conduction; Efficacy; Life expectancy expected to exceed one year with a good functional status; QRS morphology : NICD according to the AHA/ACCF/HRS Recommendations (non-LBBB and non-RBBB):; QRS duration > 130 ms
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- CRT-D or CRT-P ON (Experimental): This is a pilot, prospective, controlled, two-parallel arm, randomized, double-blind design and multicentric clinical trial comparing a CRT-D or CRT-P ON group vs. CRT-D or CRT-P OFF group in HF with reduced ejection fraction patients with NICD.
  Interventions: Other: CRT implantation
- CRT-D or CRT-P OFF (Other): This is a pilot, prospective, controlled, two-parallel arm, randomized, double-blind design and multicentric clinical trial comparing a CRT-D or CRT-P ON group vs. CRT-D or CRT-P OFF group in HF with reduced ejection fraction patients with NICD.
  Interventions: Other: CRT implantation

INTERVENTIONS:
Other: CRT implantation

SUMMARY:
The aim of the NICD-CRT study is to assess whether CRT may be clinically beneficial in HF patients with NICD and reduced ejection fraction on 12-month HF status.

In effect, the effectiveness of cardiac resynchronization therapy in heart failure (HF) with reduced ejection fraction patients with non specific intraventricular conduction delay (NICD) has never been confirmed even if it is recommended.

At the moment, no dedicated study has already been performed to assess the benefit of CRT in patients with NICD. Results from CRT therapy are contradictory in this patient group and have only been obtained from subgroup analysis. Some of them don't show clinical benefit but others show a benefit in term of an end-diastolic and/or end-systolic left ventricular volume (decrease of the size and the volumes of left ventricule).

The AHA/ACCF guidelines, published in 2005 and updated in 2009, considered only QRS duration (≥120 ms) for the indication of CRT implantation, without any consideration for the type of conduction disorder (i.e. LBBB vs. non-LBBB), current updated 2012 ACCF/AHA/HRS guidelines, consider QRS morphology (i.e. LBBB) as the first step for CRT candidate selection in addition to QRS duration (>150 ms). Indications for resynchronization have been restricted since indication of CRT in non-LBBB patients (e.g. NICD) is only a class IIa (>150 ms, only in NYHA III and ambulatory IV; level of evidence A). The same modifications have been applied between 2011 and 2013 in the European guidelines. None is known about patients with NICD and QRS > 130 ms.

DETAILED DESCRIPTION:
This is a pilot, prospective, controlled, two-parallel arm, randomized, double-blind design and multicentric clinical trial comparing a CRT-D or CRT-P ON group vs. CRT-D or CRT-P OFF group in HF with reduced ejection fraction patients with NICD.

• Patients will be included in thirteen sites in France(Clermont-Ferrand University Hospital, Côte Basque Hospital, Bordeaux University Hospital, Saint-Augustin Clinic, Limoges University Hospital, Grenoble University Hospital, Nantes University Hospital, Nantes New Clinic, Rennes University Hospital, Saint-Etienne University Hospital, Tours University Hospital, Toulouse University Hospital, Georges Pompidou European Hospital) and two sites in the Netherlands (Maastricht University Hospital and Radboud University Medical Center)

1. At baseline a preimplantation evaluation is performed: clinical examination, ECG, six minute walk test, biology analysis, quality of life assessment, echocardiography, peak oxygen consumption.
2. At 6 months, evaluation of efficacy which is the secondary assessment criteria:

   * Quality of life: Minnesota Living With Heart Failure Questionnary: MLWHFQ) : improvement of at least 20 points
   * Functionnal capacity :

     * NYHA classification reduction ≥ 1 class,
     * 6-minute walk test improvement of at least 10 % in distance,
     * Peak oxygen consumption increased by 1.0 ml/kg/minNYHA response to CRT is the primary endpoint. It is a composite primary endpoint, including modification of: Quality of Life Score (MINNESOTA scale), NYHA functional status , 6-minute walk test and volume of the left ventricle.
   * Percentage of hospitalizations for HF, for cardiovascular reasons and for all causes Decrease >15% in end-diastolic and/or end-systolic volumes of the left ventricle.
3. At 12 months, comparison of the proportion of improved, unchanged and worsend patients (Packer Score) in both group which is the primary endpoint and new evaluation of the CRT efficacy (same as 6 months)and comparison of the death and percentage of hospitalization in both group which is the primary endpoint.

ELIGIBILITY:
Inclusion criteria :

* Patients over 18 years' old
* NYHA class II to IV ambulatory
* QRS duration > 130 ms
* Patients with sinus rhythm
* LVEF < 35%
* QRS morphology: NICD according to the AHA/ACCF/HRS Recommendations (non-LBBB and non-RBBB):

  * Not broad notched or slurred R wave in leads I, aVL, V5 and V6;
  * Presence of a Q wave in leads I, V5, V6;
  * No rsr', rsR' or rSR' pattern in leads V1 or V2.
* Life expectancy expected to exceed one year with a good functional status
* Optimal pharmacological therapy of heart failure according to clinician

Non inclusion criteria :

* Inability to understand nor decline the study,
* Impaired mobility,
* Unable to fill out questionnaire independently,
* Patients with permanent atrial fibrillation,
* Pregnant women,
* Dependant adult,
* Patients minor,
* Life expectancy < 1 year due to other causes than HF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Composite of 2 clinical endpoints combined (12 months all-cause deaths and percentage of hospitalizations for HF at 12 months) combined using an average z-score. | at 12 months
  According to z-score

SECONDARY OUTCOMES:
Evaluation of efficacy, analysis of 12- month deaths | at 6 and 12 months
  HF, cardiovascular and all causes deaths
Evaluation of efficacy, analysis of - Quality-of-life questionnaires | at 6 and 12 months
  Minnesota Living With Heart Failure Questionnaire: MLWHFQ): improvement of at least 20 points
Evaluation of efficacy, analysis of Functional capacity | at 6 and 12 months
  NYHA classification reduction ≥ 1 class, 6-minute walk test improvement of at least 10 % in distance, Peak oxygen consumption increased by 1.0 ml/kg/min
Evaluation of efficacy, analysis of Percentage of hospitalizations for HF | at 6 and 12 months
Evaluation of efficacy, analysis of left ventricule volume by echocardiography transthoracic | at 6 and 12 months
  Decrease >15% in end-diastolic and/or end-systolic volumes of the left ventricle
Evaluation of efficacy, Packer score | at 6 and 12 months
  The proportion of improved, unchanged and worsened patients in both groups. Patients are considered improved if at the final visit they experienced a favorable change in NYHA functional class or in the patient global assessment (or both) of a prespecified magnitude but did not experience any major adverse clinical events during the course of the trial.
  Patients are considered worse if they experienced a major clinical event during the planned duration of double-blind treatment or reported worsening of their NYHA class or global assessment at the final visit.
  Patients are considered unchanged if they are neither improved nor worse.

CONTACTS AND LOCATIONS:
Overall Officials: Romain ESCHALIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Eschalier R, Ploux S, Pereira B, Clementy N, Da Costa A, Defaye P, Garrigue S, Gourraud JB, Gras D, Guy-Moyat B, Leclercq C, Mondoly P, Bordachar P. Assessment of cardiac resynchronisation therapy in patients with wide QRS and non-specific intraventricular conduction delay: rationale and design of the multicentre randomised NICD-CRT study. BMJ Open. 2016 Nov 11;6(11):e012383. doi: 10.1136/bmjopen-2016-012383. PMID 27836874